CLINICAL TRIAL: NCT02674685
Title: VFEND SPECIAL INVESTIGATION FOR PROPHYLAXIS
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A1501106
Record Dates: First submitted 2016-02-03; First posted 2016-02-04 (Estimated); Results first posted 2020-07-23 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-03

CONDITIONS: Fungal Infection
MeSH Terms: conditions — Mycoses

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Examine the safety and effectiveness of Vfend [voriconazole] for prophylaxix use under general clinical practices.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing HSCT (Hematopoietic Stem Cell Transplantation).

Exclusion Criteria:

* Patients who have been previously enrolled in this study.

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The subjects who have been treated with voriconazole for prophylaxis of invasive fungal infections in patients undergoing HSCT (Hematopoietic Stem Cell Transplantation)
Sampling Method: Probability Sample
Enrollment: 241 (Actual)
Dates: Start 2016-03-11 (Actual); Primary Completion 2019-07-03 (Actual); Study Completion 2019-07-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=A1501106

RESULTS

PARTICIPANT FLOW:
Groups:
- VFEND (Voriconazole): Participants who received VFEND as indicated in the approved local product document were observed for a period of 3 years at maximum. The dosage can be adjusted as per physician's discretion.
Period: Overall Study
Arm/Group | VFEND (Voriconazole)
Started | 241 (The number is same as participants enrolled.)
Completed | 237
Not Completed | 4
Not completed — Withdrawal by Subject | 4

BASELINE CHARACTERISTICS:
Population: A total of 237 participants completed this study. Of the 237 participants, 4 participants were excluded from the safety analysis set due to the following reasons: Protocol violation (registration violation, 3; contract violation/deficiency, 1)
Arm/Group | VFEND (Voriconazole)
Number analyzed (Participants) | 233
Age, Customized [Number; unit: Participants]
  <15 years | 79
  ≥15 and <65 years | 128
  ≥65 years | 26
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 96
  Male | 137
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Reason for Use [Number; unit: Participants] — Primary prophylaxis: Prophylaxis in participants without history of fungal infection. Secondary prophylaxis: Prophylaxis in participants with history of fungal infection.
  Participants
    Primary prophylaxis | 216
    Secondary prophylaxis | 16
    Others | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Drug Reactions
Description: An adverse drug reaction (ADR) was any untoward medical occurrence attributed to VFEND in a participant who received VFEND. A serious ADR was an ADR resulting in any of the following outcomes or deemed significant for any other reason: death; life-threatening experience (immediate risk of dying); initial or prolonged inpatient hospitalization; persistent or significant disability/incapacity; congenital anomaly. Relatedness to VFEND was assessed by the physician.
Time Frame: Maximum 3 years
Population: The safety analysis set comprised of participants who satisfied the inclusion criteria and had received VFEND at least once.
Measure: Number; unit: Participants
Arm/Group | VFEND (Voriconazole)
Number analyzed (Participants) | 233
Participants
  ADR | 62
  Serious ADR | 5

2. Secondary Outcome: Number of Participants With Adverse Drug Reactions Not Expected From the Approved Local Product Document (Unknown Adverse Drug Reactions)
Description: An adverse drug reaction (ADR) was any untoward medical occurrence attributed to VFEND in a participant who received VFEND. Expectedness of the adverse event was determined according to the Japanese package insert. Relatedness to VFEND was assessed by the physician.
Time Frame: Maximum 3 years
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | VFEND (Voriconazole)
Number analyzed (Participants) | 233
Participants | 6

3. Secondary Outcome: Proportion of Participants With Adverse Drug Reactions by Age
Description: An adverse drug reaction (ADR) was any untoward medical occurrence attributed to VFEND in a participant who received VFEND. Relatedness to VFEND was assessed by the physician. Participants with ADRs were counted by age (<15 years, ≥15 years) to assess whether it was a risk factor for the occurrence of ADRs.
Time Frame: Maximum 3 years
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | VFEND (Voriconazole)
Number analyzed (Participants) | 233
Percentage of Participants
  <15 years: number analyzed (Participants) | 79
  <15 years | 20.25 [12.043 to 30.796]
  ≥15 years: number analyzed (Participants) | 154
  ≥15 years | 29.87 [22.770 to 37.763]

4. Secondary Outcome: Proportion of Participants With Adverse Drug Reactions by Reason for Use
Description: An adverse drug reaction (ADR) was any untoward medical occurrence attributed to VFEND in a participant who received VFEND. Relatedness to VFEND was assessed by the physician. Participants with ADRs were counted by reason for use to assess whether it was a risk factor for the occurrence of ADRs.
Time Frame: Maximum 3 years
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | VFEND (Voriconazole)
Number analyzed (Participants) | 233
Percentage of Participants
  Primary prophylaxis: number analyzed (Participants) | 216
  Primary prophylaxis | 26.39 [20.641 to 32.797]
  Secondary prophylaxis: number analyzed (Participants) | 16
  Secondary prophylaxis | 31.25 [11.017 to 58.662]
  Others: number analyzed (Participants) | 1
  Others | 0.00 [0.000 to 97.500]

5. Secondary Outcome: Proportion of Participants With Adverse Drug Reactions by Long-term Use
Description: An adverse drug reaction (ADR) was any untoward medical occurrence attributed to VFEND in a participant who received VFEND. Relatedness to VFEND was assessed by the physician. Participants with ADRs were counted by long-term use to assess whether it was a risk factor for the occurrence of ADRs.
Time Frame: Maximum 3 years
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | VFEND (Voriconazole)
Number analyzed (Participants) | 233
Percentage of Participants
  <180 days: number analyzed (Participants) | 171
  <180 days | 24.56 [18.311 to 31.715]
  ≥180 days: number analyzed (Participants) | 62
  ≥180 days | 32.26 [20.940 to 45.336]

6. Secondary Outcome: Proportion of Participants Who Developed Invasive Fungal Infections (IFI Rate)
Description: IFI rate, which was defined as the percentage of participants who developed invasive fungal infections over the total number of assessable effectiveness analysis population, was presented along with the corresponding 2-sided 95% CI. Presence or absence of invasive fungal infections was judged as "without onset," "with onset," or "indeterminate" by the physician. In case of "with onset," it was classified as proven diagnosis, probable diagnosis, or possible case according to the diagnostic criteria of the European Organization for Research and Treatment of Cancer/Mycoses Study Group (EORTC/MSG). Participants judged as proven diagnosis or probable diagnosis were counted as those who developed invasive fungal infections for the calculation of IFI rate.
Time Frame: Maximum 3 years
Population: The efficacy analysis set (EAS) comprised of participants in the safety analysis set for whom the presence/absence of invasive fungal infections has been evaluated, excluding those with no information on effectiveness or non-target disease. The EAS was 199 participants. Those assessed as "indeterminate (n=1)" was excluded from the calculation.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | VFEND (Voriconazole)
Number analyzed (Participants) | 198
Percentage of Participants | 1.5 [0.31 to 4.36]

7. Secondary Outcome: Proportion of Participants Who Developed Invasive Fungal Infections (IFI Rate) by Age
Description: IFI rate, which was defined as the percentage of participants who developed invasive fungal infections over the total number of assessable effectiveness analysis population, was presented along with the corresponding 2-sided 95% CI. Presence or absence of invasive fungal infections was judged as "without onset," "with onset," or "indeterminate" by the physician. In case of "with onset," it was classified as proven diagnosis, probable diagnosis, or possible case according to the diagnostic criteria of the European Organization for Research and Treatment of Cancer/Mycoses Study Group (EORTC/MSG). Participants judged as proven diagnosis or probable diagnosis were counted as those who developed invasive fungal infections for the calculation of IFI rate. Participants who developed invasive fungal infections were counted by age (<15 years, ≥15 years) to assess whether it contributes to the clinical effectiveness.
Time Frame: Maximum 3 years
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | VFEND (Voriconazole)
Number analyzed (Participants) | 198
Percentage of Participants
  <15 years: number analyzed (Participants) | 68
  <15 years | 1.5 [0.04 to 7.92]
  ≥15 years: number analyzed (Participants) | 130
  ≥15 years | 1.5 [0.19 to 5.45]

8. Secondary Outcome: Proportion of Participants Who Developed Invasive Fungal Infections (IFI Rate) by Reason for Use
Description: IFI rate, which was defined as the percentage of participants who developed invasive fungal infections over the total number of assessable effectiveness analysis population, was presented along with the corresponding 2-sided 95% CI. Presence or absence of invasive fungal infections was judged as "without onset," "with onset," or "indeterminate" by the physician. In case of "with onset," it was classified as proven diagnosis, probable diagnosis, or possible case according to the diagnostic criteria of the European Organization for Research and Treatment of Cancer/Mycoses Study Group (EORTC/MSG). Participants judged as proven diagnosis or probable diagnosis were counted as those who developed invasive fungal infections for the calculation of IFI rate. Participants who developed invasive fungal infections were counted by reason for use to assess whether it contributes to the clinical effectiveness.
Time Frame: Maximum 3 years
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | VFEND (Voriconazole)
Number analyzed (Participants) | 198
Percentage of Participants
  Primary prophylaxis: number analyzed (Participants) | 184
  Primary prophylaxis | 1.1 [0.13 to 3.87]
  Secondary prophylaxis: number analyzed (Participants) | 14
  Secondary prophylaxis | 7.1 [0.18 to 33.87]

9. Secondary Outcome: Proportion of Participants With Successful Prophylaxis of Invasive Fungal Infections (Success Rate)
Description: Success rate, which was defined as the percentage of participants with successful prophylaxis of invasive fungal infections over the total number of assessable effectiveness analysis population, was presented along with the corresponding 2-sided 95% CI. Presence or absence of invasive fungal infections was judged as "without onset," "with onset," or "indeterminate" by the physician, and participants judged as "without onset" were counted as those with successful prophylaxis of invasive fungal infections for the calculation of success rate.
Time Frame: Maximum 3 years
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | VFEND (Voriconazole)
Number analyzed (Participants) | 198
Percentage of Participants | 97.5 [94.21 to 99.18]

10. Secondary Outcome: Proportion of Participants With Successful Prophylaxis of Invasive Fungal Infections (Success Rate) by Age
Description: Success rate, which was defined as the percentage of participants with successful prophylaxis of invasive fungal infections over the total number of assessable effectiveness analysis population, was presented along with the corresponding 2-sided 95% CI. Presence or absence of invasive fungal infections was judged as "without onset," "with onset," or "indeterminate" by the physician, and participants judged as "without onset" were counted as those with successful prophylaxis of invasive fungal infections for the calculation of success rate. Participants with successful prophylaxis of invasive fungal infections were counted by age (<15 years, ≥15 years) to assess whether it contributes to the clinical effectiveness.
Time Frame: Maximum 3 years
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | VFEND (Voriconazole)
Number analyzed (Participants) | 198
Percentage of Participants
  <15 years: number analyzed (Participants) | 68
  <15 years | 98.5 [92.08 to 99.96]
  ≥15 years: number analyzed (Participants) | 130
  ≥15 years | 96.9 [92.31 to 99.16]

11. Secondary Outcome: Proportion of Participants With Successful Prophylaxis of Invasive Fungal Infections (Success Rate) by Reason for Use
Description: Success rate, which was defined as the percentage of participants with successful prophylaxis of invasive fungal infections over the total number of assessable effectiveness analysis population, was presented along with the corresponding 2-sided 95% CI. Presence or absence of invasive fungal infections was judged as "without onset," "with onset," or "indeterminate" by the physician, and participants judged as "without onset" were counted as those with successful prophylaxis of invasive fungal infections for the calculation of success rate. Participants with successful prophylaxis of invasive fungal infections were counted by reason for use to assess whether it contributes to the clinical effectiveness.
Time Frame: Maximum 3 years
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | VFEND (Voriconazole)
Number analyzed (Participants) | 198
Percentage of Participants
  Primary prophylaxis: number analyzed (Participants) | 184
  Primary prophylaxis | 97.8 [94.53 to 99.40]
  Secondary prophylaxis: number analyzed (Participants) | 14
  Secondary prophylaxis | 92.9 [66.13 to 99.82]

ADVERSE EVENTS:
Time Frame: 3 years at Maximum
Description: The frequency of adverse events. The same event may appear as both an adverse event and a serious adverse event. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another participant, or one participant may have experienced both serious and non-serious events during the study.
Arm/Group | VFEND (Voriconazole)
All-Cause Mortality (participants affected / at risk) | 19/233
Serious Adverse Events (participants affected / at risk) | 60/233
Other Adverse Events (participants affected / at risk) | 153/233
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | VFEND (Voriconazole) (N=233)
Adenovirus infection (Infections and infestations) | 1
Pneumonia influenzal (Infections and infestations) | 1
Cytomegalovirus viraemia (Infections and infestations) | 1
Staphylococcal sepsis (Infections and infestations) | 1
Herpes virus infection (Infections and infestations) | 1
Meningoencephalitis herpetic (Infections and infestations) | 1
Bacteraemia (Infections and infestations) | 1
Psoas abscess (Infections and infestations) | 1
Tooth infection (Infections and infestations) | 1
Systemic candida (Infections and infestations) | 1
Systemic mycosis (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 3
Lung abscess (Infections and infestations) | 1
Acute lymphocytic leukaemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Chronic myeloid leukaemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Anaemia (Blood and lymphatic system disorders) | 1
Bone marrow failure (Blood and lymphatic system disorders) | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 5
Immune thrombocytopenic purpura (Blood and lymphatic system disorders) | 1
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 1
Acute graft versus host disease (Immune system disorders) | 3
Acute graft versus host disease in intestine (Immune system disorders) | 1
Acute graft versus host disease in liver (Immune system disorders) | 1
Cytokine storm (Immune system disorders) | 1
Engraftment syndrome (Immune system disorders) | 1
Graft versus host disease (Immune system disorders) | 12
Graft versus host disease in lung (Immune system disorders) | 2
Primary amyloidosis (Immune system disorders) | 1
Tumour lysis syndrome (Metabolism and nutrition disorders) | 2
Cerebrovascular accident (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Parkinsonism (Nervous system disorders) | 1
Arrhythmia (Cardiac disorders) | 1
Cardiac failure (Cardiac disorders) | 1
Cardiac failure acute (Cardiac disorders) | 1
Cardiac failure chronic (Cardiac disorders) | 1
Shock (Vascular disorders) | 1
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 1
Idiopathic pneumonia syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Pancreatitis acute (Gastrointestinal disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 1
Hepatic function abnormal (Hepatobiliary disorders) | 1
Hepatitis acute (Hepatobiliary disorders) | 1
Venoocclusive liver disease (Hepatobiliary disorders) | 2
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 2
Nephrotic syndrome (Renal and urinary disorders) | 1
Renal disorder (Renal and urinary disorders) | 1
Renal failure (Renal and urinary disorders) | 1
Renal impairment (Renal and urinary disorders) | 4
Generalised oedema (General disorders) | 1
Mucosal inflammation (General disorders) | 1
Multiple organ dysfunction syndrome (General disorders) | 1
Aspartate aminotransferase increased (Investigations) | 1
Blood bilirubin increased (Investigations) | 3
Blood creatinine increased (Investigations) | 2
Blood urea increased (Investigations) | 1
Neutrophil count decreased (Investigations) | 3
Platelet count decreased (Investigations) | 2
Engraft failure (Injury, poisoning and procedural complications) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | VFEND (Voriconazole) (N=233)
Anaemia (Blood and lymphatic system disorders) | 8
Bone marrow failure (Blood and lymphatic system disorders) | 4
Eosinophilia (Blood and lymphatic system disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 33
Leukopenia (Blood and lymphatic system disorders) | 5
Neutropenia (Blood and lymphatic system disorders) | 8
Pancytopenia (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 10
Photophobia (Eye disorders) | 9
Photopsia (Eye disorders) | 1
Visual impairment (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 3
Dyschezia (Gastrointestinal disorders) | 1
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1
Gastrointestinal mucosal disorder (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 5
Oral disorder (Gastrointestinal disorders) | 4
Stomatitis (Gastrointestinal disorders) | 6
Vomiting (Gastrointestinal disorders) | 2
Mucosal disorder (General disorders) | 1
Oedema (General disorders) | 1
Pyrexia (General disorders) | 2
Bile duct stone (Hepatobiliary disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 1
Cholelithiasis (Hepatobiliary disorders) | 1
Cholestasis (Hepatobiliary disorders) | 1
Hepatic function abnormal (Hepatobiliary disorders) | 8
Hepatotoxicity (Hepatobiliary disorders) | 2
Liver disorder (Hepatobiliary disorders) | 14
Venoocclusive liver disease (Hepatobiliary disorders) | 3
Acute graft versus host disease (Immune system disorders) | 1
Acute graft versus host disease in intestine (Immune system disorders) | 1
Acute graft versus host disease in skin (Immune system disorders) | 4
Anaphylactic reaction (Immune system disorders) | 1
Engraftment syndrome (Immune system disorders) | 7
Graft versus host disease (Immune system disorders) | 31
Graft versus host disease in liver (Immune system disorders) | 1
Graft versus host disease in skin (Immune system disorders) | 5
Hypogammaglobulinaemia (Immune system disorders) | 1
Aspergillus infection (Infections and infestations) | 1
Bacterial infection (Infections and infestations) | 1
Candida infection (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Cytomegalovirus infection (Infections and infestations) | 3
Cytomegalovirus viraemia (Infections and infestations) | 10
Fungal infection (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 1
Oesophageal candidiasis (Infections and infestations) | 1
Oral herpes (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Skin infection (Infections and infestations) | 1
Tongue fungal infection (Infections and infestations) | 1
Alanine aminotransferase decreased (Investigations) | 1
Alanine aminotransferase increased (Investigations) | 24
Aspartate aminotransferase increased (Investigations) | 23
Blood alkaline phosphatase increased (Investigations) | 19
Blood beta-D-glucan increased (Investigations) | 1
Blood bilirubin increased (Investigations) | 5
Blood creatinine increased (Investigations) | 5
Blood lactate dehydrogenase increased (Investigations) | 2
Blood pressure increased (Investigations) | 1
Blood urea increased (Investigations) | 4
Brain natriuretic peptide increased (Investigations) | 1
C-reactive protein increased (Investigations) | 9
Drug level increased (Investigations) | 1
Electrocardiogram QT prolonged (Investigations) | 1
Gamma-glutamyltransferase increased (Investigations) | 30
International normalised ratio increased (Investigations) | 1
Neutrophil count decreased (Investigations) | 4
Platelet count decreased (Investigations) | 12
Serum ferritin increased (Investigations) | 1
Transaminases increased (Investigations) | 2
White blood cell count decreased (Investigations) | 12
White blood cell count increased (Investigations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 2
Diabetes mellitus (Metabolism and nutrition disorders) | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1
Hypochloraemia (Metabolism and nutrition disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1
Steroid diabetes (Metabolism and nutrition disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Bone formation increased (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Myopathy (Musculoskeletal and connective tissue disorders) | 1
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Headache (Nervous system disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1
Delirium (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 1
Hallucination, auditory (Psychiatric disorders) | 1
Hallucination, visual (Psychiatric disorders) | 2
Insomnia (Psychiatric disorders) | 1
Azotaemia (Renal and urinary disorders) | 1
Cystitis haemorrhagic (Renal and urinary disorders) | 1
Hydronephrosis (Renal and urinary disorders) | 1
Renal impairment (Renal and urinary disorders) | 5
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1
Drug eruption (Skin and subcutaneous tissue disorders) | 2
Pruritus (Skin and subcutaneous tissue disorders) | 2
Rash (Skin and subcutaneous tissue disorders) | 4
Hypertension (Vascular disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2015-09-02): https://cdn.clinicaltrials.gov/large-docs/85/NCT02674685/Prot_001.pdf
  • Statistical Analysis Plan (2019-06-10): https://cdn.clinicaltrials.gov/large-docs/85/NCT02674685/SAP_000.pdf